CLINICAL TRIAL: NCT00624520
Title: Effectiveness of Mental Stress Reduction in Defibrillator Patients
Brief Title: Mental Stress Reduction in Defibrillator Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Exhaustion of subject population pool, greater than expected drop-out rates . Data analysis approved by DMC for study completions
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-008-07F
Record Dates: First submitted 2008-02-14; First posted 2008-02-27 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Cardiomyopathy, Dilated; Arrhythmia; Anger; Stress
Keywords: Stress, Psychological; Tachycardia, Ventricular; Defibrillators, Implantable; Death, Sudden Cardiac; Cognitive Therapy; Anger
MeSH Terms: conditions — Cardiomyopathy, Dilated; Arrhythmias, Cardiac; Stress, Psychological; Tachycardia, Ventricular; Death, Sudden, Cardiac | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Stress Management (Active Comparator): 10 week program of Cognitive Behavioral Stress Management (CBSM) group sessions
  Interventions: Behavioral: Cognitive Behavioral Stress Management (CBSM)
- Patient Education (Active Comparator): 10 week program of once weekly Patient Education group sessions
  Interventions: Other: Patient Education

INTERVENTIONS:
Behavioral: Cognitive Behavioral Stress Management (CBSM) — 10 week program of weekly CBSM therapy group sessions
  Arms: Cognitive Behavioral Stress Management
Other: Patient Education — 10 week program of "Patient Education" group sessions, involving presentations of educational materials relating to heart disease.
  Arms: Patient Education

SUMMARY:
The purpose of this study is to assess the effectiveness of a 10 week program of Stress Management versus control Patient Education sessions on cardiac responses to mental stress in veterans with Implantable Cardioverter-Defibrillators

DETAILED DESCRIPTION:
The study is a randomized controlled small clinical trial designed to determine whether a 10-week program of group cognitive-behavioral stress management (CBSM) versus a control "Patient Education" program can improve hemodynamic responses to mental stress testing in patients with Implantable Cardioverter Defibrillators. Comparison will be made between groups of heart rate and blood pressure responses to mental arithmetic and anger-recall mental stress, psychometric profiles, arrhythmia frequency and implantable cardioverter defibrillator firings before, immediately and up to 6 months after intervention. If benefit of CBSM is proven, study findings could lead to wider use of stress management programs, with increased life expectancy for implantable cardioverter-defibrillator patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >21 years,
* ICD Implantation,
* > 3 months following ICD implantation,
* willingness to give informed consent

Exclusion Criteria:

* Episodes within prior 3 months of: acute coronary syndrome, myocardial infraction, Coronary Artery By-pass Graft surgery, percutaneous coronary intervention, hospital admission any cause,
* severe mental illness,
* life expectancy < 1 year,
* hyperkalemia,
* hypokalemia,
* hypomagnesemia,
* hypermagnesemia,
* unwillingness to give informed consent

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Russell, MD PhD, Principal Investigator — Wlliam S. Middleton Memorial Veterans Hospital, Madison
Locations (2):
- United States (2):
  - Wlliam S. Middleton Memorial Veterans Hospital, Madison, Madison, Wisconsin
  - Zablocki VA Medical Center, Milwaukee, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Russell DC, Smith TL, Krahn DD, Graskamp P, Singh D, Kolden GG, Sigmund H, Zhang Z. Effects of Cognitive Behavioral Stress Management on Negative Mood and Cardiac Autonomic Activity in ICD Recipients. Pacing Clin Electrophysiol. 2015 Aug;38(8):951-65. doi: 10.1111/pace.12668. Epub 2015 Jun 20. PMID 26010524

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment commenced October 2009, completed December 2011 Recruitment from Cardiology Clinics W S Middleton Veterans Hospital, Madison, and Zablocki VA Medical Center, Milwaukee
Pre-assignment Details: Some enrolled participants were excluded from the trial if determined to have severe mental illness after administration of an SCID-I questionnaire and/or interview by a clinical psychologist. Others were excluded as drop-outs due to travel issues, weather, family issues, and illness. 2 subjects died before group assignment.
Period: Overall Study
Arm/Group | Cognitive Behavioral Stress Management | Patient Education
Started | 56 | 47
Completed | 44 | 39
Not Completed | 12 | 8
Not completed — Withdrawal by Subject | 12 | 7
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects randomized , including drop-outs before commencement of intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Stress Management | Patient Education | Total
Number analyzed (Participants) | 56 | 47 | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (9.0) | 66.2 (8.6) | 65.7 (8.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 23 | 55
  >=65 years | 24 | 24 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 56 | 46 | 102
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 51 | 41 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 56 | 45 | 101
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Madison and Milwaukee study sites, US
  participants
    United States | 56 | 47 | 103

OUTCOME MEASURES:

1. Primary Outcome: Mental Stress Induced Elevation in "Double Product" by Math Stress Task
Description: Maximum Mental Stress induced elevation in "Double Product" , (equal to Heart Rate , beats/minute, x Systolic Arterial Blood Pressure, mmHg), following serial heart rate and blood pressure measurements during mental stress task of mental arithmetic (serial subtraction). Heart rate and blood pressure responses were recorded at 2.5 minute intervals before , during, and after each test using a Philips automated blood pressure recording device. The math task was applied for 10 minutes, with 10 minutes recovery time. An average of 3 measurements was taken as baseline prior to stress tasks. Stress induced double product elevations were measured as the difference between baseline and maximal values in units of mmHg.beats/minute. Higher values represent a greater mental stress induced effect, and lower values, a lower effect.
Time Frame: Immediate to 6 months post intervention
Population: Response to Mental Stress by Math Stress Task.
Measure: Mean (Standard Error); unit: mmHg x beats/min
Arm/Group | Cognitive Behavioral Stress Management | Patient Education
Number analyzed (Participants) | 43 | 38
mmHg x beats/min
  6 months post | 1693 (343) | 1137 (228)
  3 months post | 1399 (201) | 1063 (158)
  Immediate post | 1514 (246) | 1538 (224)
Statistical Analysis 1: Comparison: Cognitive Behavioral Stress Management vs Patient Education; Initial sample size calculation, based on previous published data of effects sizes of anger stress management on heart rate and blood pressure responses in a veteran population, indicated a study population of 138 patients should detect a reduction in "Double Product" response to mental stress following psychological intervention, with over 90% power, assuming 20% drop-out rate; Test type: Superiority or Other; p = 0.18, ANOVA — Statistical Analysis presented for comparison groups Cognitive Behavioral Stress Management vs. Patient Education at 6 months post; Mean Difference (Final Values) = 891

2. Secondary Outcome: State Anger
Description: Psychosocial score of negative mood derived from self-report questionnaires. Scale range was 15-45. Lower values represent better outcome, and higher values represent worse outcome..
Time Frame: Immediate post intervention
Population: Serial psychometric scores up to 6 months post intervention Reduced numbers of participants analyzed reflect drop-outs or failure to fully complete questionnaires during follow-up, with inclusion only of participants having accurate and appropriate data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Stress Management | Patient Education
Number analyzed (Participants) | 39 | 36
units on a scale | 16 (2) | 19 (7)
Statistical Analysis 1: Comparison: Cognitive Behavioral Stress Management vs Patient Education; Test type: Superiority or Other; p = 0.02, ANOVA; Mean Difference (Final Values) = 3

3. Secondary Outcome: Tension/Anxiety
Description: Psychometric score by self-report questionnaire Scale range is 3-29. Lower values represent better outcome, and higher values represent worse outcome..
Time Frame: Immediate post intervention
Population: Immediate post intervention Reduced numbers of participants analyzed reflect drop-outs or failure to fully complete questionnaires during follow-up, with inclusion only of participants having accurate and appropriate data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Stress Management | Patient Education
Number analyzed (Participants) | 39 | 38
units on a scale | 8 (4) | 12 (7)
Statistical Analysis 1: Comparison: Cognitive Behavioral Stress Management vs Patient Education; Test type: Superiority or Other; p = 0.003, ANOVA; Mean Difference (Final Values) = -4

4. Secondary Outcome: Perceived Stress
Description: Psychometric score from self-report questionnaire Scale range is 2-27. Lower values represent better outcome, and higher values represent worse outcome..
Time Frame: Immediate post intervention
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Stress Management | Patient Education
Number analyzed (Participants) | 39 | 38
units on a scale | 10 (6) | 14 (8)
Statistical Analysis 1: Comparison: Cognitive Behavioral Stress Management vs Patient Education; Test type: Superiority or Other; p = 0.011, ANOVA; Mean Difference (Final Values) = -4

5. Secondary Outcome: Depression/Dejection
Description: Psychometric score from self-report questionnaire Scale range is 9 to 60. Lower values represent better outcome, and higher values represent worse outcome..
Time Frame: 3 months post intervention
Population: 3 months post intervention Reduced numbers of participants analyzed reflect drop-outs or failure to fully complete questionnaires during follow-up,with inclusion only of participants having accurate and appropriate data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Stress Management | Patient Education
Number analyzed (Participants) | 38 | 38
units on a scale | 20 (6) | 24 (11)
Statistical Analysis 1: Comparison: Cognitive Behavioral Stress Management vs Patient Education; Test type: Superiority or Other; p = 0.048, ANOVA; Mean Difference (Final Values) = -4

6. Secondary Outcome: Low Frequency Heart Rate Variability
Description: Heart Rate Variability measure of cardiac autonomic activity, believed to reflect a combination of cardiac sympathetic and parasympathetic activity.
  Data are derived from ambulatory ECG recordings during serial mental stress testing (math and anger-recall tasks) using a General Electric MARS Holter analysis system. Time series are created from beat-to-beat intervals, from which frequency domain measures are calculated. Low frequency heart rate variability correlates with cardiac sympathetic and parasympathetic activity. Increased sympathetic activity and/or decreased parasympathetic activity occur in this study population at high risk for cardiac arrhythmia. Normalized units are used, reflecting percentage of total frequency power.
Time Frame: 6 months post intervention
Population: 6 months post intervention, from ECG recordings during mental stress tasks Reduced numbers of participants analyzed reflect drop-outs or non-diagnostic recordings for HRV analyses during follow-up, with inclusion only of participants having accurate and appropriate data.
Measure: Mean (Standard Deviation); unit: percentage of spectral power
Arm/Group | Cognitive Behavioral Stress Management | Patient Education
Number analyzed (Participants) | 17 | 23
percentage of spectral power | 59 (19) | 70 (21)
Statistical Analysis 1: Comparison: Cognitive Behavioral Stress Management vs Patient Education; Test type: Superiority or Other; p = 0.01, ANOVA; Mean Difference (Final Values) = -11

7. Secondary Outcome: High Frequency Heart Rate Variability
Description: Heart Rate Variability measure of Cardiac Parasympathetic activity. Data are derived from ambulatory ECG recordings during serial mental stress testing (math and anger-recall tasks) using a General Electric MARS Holter analysis system. Time series are created from beat-to-beat intervals, from which frequency domain measures are calculated. Increased High Frequency heart rate variability correlates with increased cardiac parasympathetic activity. Normalized units are used, reflecting percentage of total frequency power.
Time Frame: 6 months post intervention
Population: Reduced participant numbers reflect drop-outs and exclusion of participants with non-diagnostic recordings for HRV analyses, with inclusion only of participants having accurate and appropriate data.
Measure: Mean (Standard Deviation); unit: percentage of spectral power
Arm/Group | Cognitive Behavioral Stress Management | Patient Education
Number analyzed (Participants) | 17 | 23
percentage of spectral power | 41 (19) | 26 (16)
Statistical Analysis 1: Comparison: Cognitive Behavioral Stress Management vs Patient Education; Test type: Superiority or Other; p = 0.01, ANOVA; Mean Difference (Final Values) = 15

8. Secondary Outcome: Low Frequency/High Frequency Ratio of Heart Rate Variability
Description: Heart Rate Variability measure of cardiac autonomic activity Data are derived from ambulatory ECG recordings during serial mental stress testing (math and anger-recall tasks) using a General Electric MARS Holter analysis system. Time series are created from beat-to-beat intervals, from which frequency domain measures are calculated. Decreased Low/High Frequency ratio reflects Increased High Frequency heart rate variability which correlates with increased cardiac parasympathetic activity, which may be beneficial in this patient population. Normalized units are used, reflecting percentage of total frequency power.
Time Frame: 6 months post intervention
Population: Reduced numbers of participants analyzed reflect drop-outs or non-diagnostic recordings for heart rate variability analyses during follow-up, with inclusion only of participants having accurate and appropriate data.
  Data are shown for Ratios of Low and High Frequency power shown above.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cognitive Behavioral Stress Management | Patient Education
Number analyzed (Participants) | 17 | 23
Ratio | 1.99 (1.47) | 4.01 (3.26)
Statistical Analysis 1: Comparison: Cognitive Behavioral Stress Management vs Patient Education; Test type: Superiority or Other; p = 0.01, ANOVA; Mean Difference (Final Values) = -2.02

9. Secondary Outcome: Cardioverter-DefibrillatorTherapies
Description: Cardioverter-Defibrillator therapies for treatment of serious ventricular arrhythmia
Time Frame: 6 months post intervention
Population: Cardioverter-defibrillator interrogation data between 3 and 6 months post intervention
Measure: Number; unit: percentage of participants
Arm/Group | Cognitive Behavioral Stress Management | Patient Education
Number analyzed (Participants) | 38 | 33
percentage of participants | 0 | 6
Statistical Analysis 1: Comparison: Cognitive Behavioral Stress Management vs Patient Education; Test type: Superiority or Other; p = 0.21, Fisher Exact

10. Primary Outcome: Mental Stress Induced Elevation in Double Product by Math Stress Task
Description: Maximum Mental Stress induced elevation in "Double Product" , DP, (equal to Heart Rate , beats/minute, x Systolic Arterial Blood Pressure, mmHg), following serial heart rate and blood pressure measurements during mental stress tasks of mental arithmetic (serial subtraction). Heart rate and blood pressure responses were recorded at 2.5 minute intervals before , during, and after each test using a Philips automated blood pressure recording device. The math task was applied for 10 minutes, with 10 minutes recovery time. An average of 3 measurements was taken as baseline prior to stress tasks. Stress induced double product elevations were measured as the difference between baseline and maximal values in units of mmHg.beats/minute. Higher values represent a greater mental stress induced effect, and lower values, a lower effect.
Time Frame: 3 months post intervention
Population: Response to mental stress by math task testing at 3 months post intervention, compared with pre-intervention. Within-group comparison is shown for matched pair data. The lower number of participants analyzed than at study entry is due to patient drop-outs during follow-up post-intervention.
Measure: Mean (Standard Error); unit: mmHg x beats/minute
Arm/Group | Cognitive Behavioral Stress Management
Number analyzed (Participants) | 36
mmHg x beats/minute
  Pre intervention | 1915 (263)
  3 months post intervention | 1399 (201)
Statistical Analysis 1: Comparison: Cognitive Behavioral Stress Management; Test type: Superiority or Other; p = 0.025, ANCOVA — P-value refers to a repeated measures within-group comparison in the CBSM group using ANCOVA with baseline DP elevation as covariate from baseline to 3 months post; Effect size (Cohen's d) = 0.38 — Range of Cohen's d for small effect is 0.20 - 0.50

11. Primary Outcome: Mental Stress Induced Elevation in "Double Product" by Anger-recall Task
Description: Maximum Mental Stress induced elevation in "Double Product" , (equal to Heart Rate , beats/minute, x Systolic Arterial Blood Pressure, mmHg), following serial heart rate and blood pressure measurements during mental stress of anger-recall task. Heart rate and blood pressure responses were recorded at 2.5 minute intervals before , during, and after each test using a Philips automated blood pressure recording device. The anger-recall test was applied for 25 minutes with 10 minutes monitoring post-test. An average of 3 measurements was taken as baseline prior to stress tasks. Stress induced double product elevations were measured as the difference between baseline and maximal values in units of mmHg.beats/minute. Higher values represent a greater mental stress induced effect, and lower values, a lower effect
Time Frame: Immediate to 6 months post intervention
Population: Response to Mental Stress by Anger-Recall Stress Task
Measure: Mean (Standard Error); unit: mmHg x beats/minute
Arm/Group | Cognitive Behavioral Stress Management | Patient Education
Number analyzed (Participants) | 44 | 39
mmHg x beats/minute
  6 months post intervention | 711 (232) | 631 (292)
  3 months post intervention | 353 (167) | 548 (308)
  Immediate post intervention | 406 (93) | 681 (244)
Statistical Analysis 1: Comparison: Cognitive Behavioral Stress Management vs Patient Education; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.81, ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 80

ADVERSE EVENTS:
Time Frame: 6 to 12 months, from enrollment to study completion
Arm/Group | Cognitive Behavioral Stress Management | Patient Education
Serious Adverse Events (participants affected / at risk) | 9/56 | 12/47
Other Adverse Events (participants affected / at risk) | 0/56 | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Stress Management (N=56) | Patient Education (N=47)
Death (Cardiac disorders) | 0 (0) | 1 (1) — Cardiomyopathy, sudden cardiac death
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0) — Includes Ablation procedures
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — Tachycardia unknown origin
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Dizziness (Cardiac disorders) | 1 (2) | 2 (2) — Includes syncope, dizziness, hypotension
Implantable Defibrillator malfunction (Cardiac disorders) | 2 (3) | 1 (1) — Includes admissions for inappropriate device firings, lead revisions
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal stricture (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Includes colonoscopy
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Carotid artery disease (Vascular disorders) | 1 (1) | 0 (0) — Includes carotid artery surgery
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — includes respiratory infection
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Includes nasal polypectomy
Cerebrovascular Disease (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of study after 12 month study extension and interim data analysis, due to high drop-out rate and exhaustion of population pool, 9 subjects short of revised target enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes